CLINICAL TRIAL: NCT00619892
Title: An 8-week, Randomized, Double-Blind, Placebo-Controlled Trial of Seroquel SR Co-administration for SSRI-Resistant, Comorbid Panic Disorder
Brief Title: A Study of Quetiapine SR (Seroquel SR) to Treat SSRI-Resistant, Comorbid Panic Disorder Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0703-22; IRUSQUET0445 (Other Grant/Funding Number: Astra Zeneca)
Record Dates: First submitted 2008-02-11; First posted 2008-02-21 (Estimated); Results first posted 2016-01-21 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2015-12

CONDITIONS: Panic Disorder
Keywords: SSRI Resistant; Seroquel SR; Seroquel XR; Panic Disorder; Comorbid Panic Disorder; Quetiapine SR; Quetiapine XR
MeSH Terms: conditions — Panic Disorder | interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Quetiapine XR (Active Comparator): Our target daily dose for quetiapine XR was 200 mg/day. The detailed quetiapine XR dosing guidelines were as follows: 50 mg 1 tab po at HS × 3 days, then, if 50 mg tolerated, increase to 50 mg 2 tabs at HS × 4 days; at the beginning of week 2, if the last dose was tolerated increase to 50 mg 3 tabs at HS × 3 days, then, if 150 mg tolerated, increase to 4 tabs at HS; at the beginning of week 3, if no efficacy & the 200 mg dose was well tolerated, increase to one 300 mg tab at HS-otherwise remain at 200 mg one tab at HS; at week 4 if still no improvement, & 300 mg was tolerable, increase to 200 mg tablet 2 at HS. From the beginning of week 5 to the end of the trial, quetiapine XR doses were held. We used quetiapine XR tablets provided by Astra Zeneca (50, 200, and 300 mg designations).
  Interventions: Drug: quetiapine XR
- Placebo (Placebo Comparator): Subjects received identical-appearing placebo tablets provided by Astra Zeneca (50, 200, and 300 mg designations).
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: quetiapine XR — Subjects will receive daily dosing at night, with a flexible dosing schedule, 50-400 mg.
  Other Names: Seroquel SR; Seroquel XR
  Arms: Quetiapine XR
Drug: placebo — Subjects will receive daily dosing at night with caplets matching the appearance of the active drug. However, caplets will not contain any active medication.
  Other Names: Astra Zeneca placebo
  Arms: Placebo

SUMMARY:
The primary objective of this study is to test the hypothesis that a SSRI plus quetiapine SR (Seroquel SR) will result in superior early (first 1-3 weeks of treatment) stabilization of panic symptoms in SSRI-resistant, comorbid Panic Disorder patients versus a SSRI plus placebo.

DETAILED DESCRIPTION:
This was a single-site, double-blind, placebo-controlled (PLAC), randomized, parallel group (2 groups), 8-week, quetiapine extended release (XR) coadministration trial. SSRI resistance was determined either historically or prospectively. Patients were randomized if they remained moderately ill (CGI-S score ≥ 4). Change in the PDSS scale total score was the primary efficacy outcome measure. Responders were identified as those with a ≥50 % decrease from their baseline PDSS score. In the early weeks of therapy, XR was flexibly and gradually titrated from 50 to 400 mg/day.

Conclusions: This proof-of-concept RCT did not support the efficacy of this treatment strategy for SSRI-resistant PD. Quetiapine XR was generally well-tolerated. Important limitations were the small sample size, and the relatively low average dose of quetiapine XR used.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Diagnosis of Panic Disorder by DSM-IV TR and confirmed by MINI plus interview
* Females and males ages 18-65 years old
* Female patients of childbearing potential must by using a reliable method of contraception and have a negative urine human chorionic gonadotropin (HCG) test at enrollment
* Able to understand and comply with the requirements of the study
* Have a CGI illness severity score = or > 4
* Patients with comorbid major depression, dysthymia or other anxiety problems are eligible to participate as well.

Exclusion criteria:

* Pregnancy or lactation
* Any DSM-IV TR Axis I disorder not mentioned in the inclusion requirements
* Suicidal or danger to self or others
* Known intolerance to quetiapine fumarate or intolerance to SSRI therapy
* Use of any of the following cytochrome P450 3A4 inhibitors in the 14 days preceding enrollment including but not limited to : ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, troleandomycin, indinavir, nelfinavir, ritonavir, fluvoxamine and saquinavir
* Use of any of the following cytochrome P450 inducers in the 14 days preceding enrollment including but not limited to : phenytoin, carbamazepine, barbiturates, rifampin, St. John's Wort, and glucocorticoids
* Administration of a depot antipsychotic injection within one dosing interval (for the depot) before randomization
* Substance or alcohol dependence at enrollment (except dependence in full remission, and except for caffeine or nicotine dependence), as defined by DSM-IV criteria
* Opiates, amphetamine, barbiturate, cocaine, cannabis, or hallucinogen abuse by DSM-IV TR criteria within 4 weeks prior to enrollment
* Medical conditions that would affect absorption, distribution, metabolism, or excretion of study treatment
* Unstable or inadequately treated medical illness (e.g. angina pectoris, hypertension) as judged by the investigator
* Involvement in the planning and conduct of the study
* Previous enrollment or randomization of treatment in the present study
* Participation in another drug trial within 4 weeks prior enrollment into this study or longer in accordance with local requirements
* A patient with a diagnosis of Type I or Type II Diabetes Mellitus (DM)
* An absolute neutrophil count (ANC) of 1.5 x 109 per liter
* A lifetime history of a pre-existing CNS/neurological disorder e.g. epilepsy, TBI, brain tumor
* Patient with severe personality disorders
* Patients who have started a new course of psychotherapy (CBT, supportive, insight-oriented) within 1 month of the screening visit
* Patients unwilling to refrain from participation in psychotherapy during the 9-week period of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2008-02; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew W. Goddard, M.D., Principal Investigator — Indiana University
Locations (1):
- University Hospital Outpatient Center, Psychiatry, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Goddard AW, Mahmud W, Medlock C, Shin YW, Shekhar A. A controlled trial of quetiapine XR coadministration treatment of SSRI-resistant panic disorder. Ann Gen Psychiatry. 2015 Sep 15;14:26. doi: 10.1186/s12991-015-0064-0. eCollection 2015. PMID 26379759

RESULTS

PARTICIPANT FLOW:
Groups:
- Quetiapine SR: quetiapine SR: Subjects will receive daily dosing at night, with a flexible dosing schedule, 50-400 mg.
Period: Overall Study
Arm/Group | Quetiapine SR | Placebo
Started | 13 | 13
Completed | 10 | 11
Not Completed | 3 | 2
Not completed — Adverse Event | 3 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Intercurrent illness | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Quetiapine: Quetiapine SR: Subjects will receive daily dosing at night, with a flexible dosing schedule, 50-400 mg.
- Total: Total of all reporting groups
Arm/Group | Quetiapine | Placebo | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 13 | 26
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.5 (9.6) | 35.5 (16.8) | 35.5 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 3 | 5 | 8
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 26
Panic Disorder Severity Scale [Mean (Standard Deviation); unit: units on a scale] — Possible range 0-28 (7 questions, each scored from 0 to 4, with higher numbers indicating more severe panic symptoms).
  Mean (Standard Deviation)
  units on a scale | 14.8 (3.6) | 13.7 (3) | 14.3 (3.3)
Clinical Global Impression-Severity Scale (CGI-S) [Mean (Standard Deviation); unit: units on a scale] — CGI-S is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, where 1 =normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; or 7 = extremely ill.
  units on a scale | 4.8 (0.8) | 4.4 (0.7) | 4.6 (0.8)
Hamilton Anxiety Rating Scale (HAM-A) [Mean (Standard Deviation); unit: units on a scale] — Hamilton Anxiety Rating Scale (HAM-A) is a questionnaire used by clinicians to rate the severity of a patient's anxiety. The scale consists of 14 items designed to assess the severity of a patient's anxiety, each of which is rated on a scale of 0 to 4, with 4 being the most severe. Total scores can range from 0 to 56.
  units on a scale | 21.2 (6.8) | 17 (5.2) | 19.1 (6.0)
Hamilton Depression Rating Scale (HAM-D) [Mean (Standard Deviation); unit: units on a scale] — The HAM-D is a questionnaire with 17 items. Each item on the questionnaire is scored on a 3 or 5 point scale. The total scores indicate levels of depression, where 0-7= normal; 8-13 = mild depression; 14-18 = moderate depression; 19-22 = severe depression; and 23 or greater = very severe depression.
  units on a scale | 14.6 (6.2) | 11.5 (5.1) | 13.1 (5.7)
Pittsburgh Sleep Quality Index (PSQI) sleep hours [Mean (Standard Deviation); unit: hours slept per night] — The PSQI sleep hours subscale is a self-reported measure of the number of hours patients slept per night over the past month.
  hours slept per night | 6.2 (1.3) | 6.7 (1.6) | 6.5 (1.5)
Pittsburgh Sleep Quality Index (PSQI) sleep quality [Mean (Standard Deviation); unit: units on a scale] — The PSQI sleep quality subscale is a self-reported measure of the patient's sleep quality over the past month, with a possible range of 0-3, where 0 = very good; 1 = fairly good; 2= fairly bad; and 3 = very bad.
  units on a scale | 2.9 (0.6) | 2.3 (0.6) | 2.6 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Total Panic Disorder Severity Scale (PDSS) Scores
Description: Possible total scores on the PDSS range from 0-28. The outcome measure represents the change, between baseline and the end of 8 weeks of treatment, in the the total PDSS scores. Lower scores indicate less severe panic disorder symptoms. A negative mean change in the scores at the end of 8 weeks represents a decrease in severity of panic disorder symptoms.
Time Frame: Baseline and the end of 8 weeks of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Quetiapine SR | Placebo
Number analyzed (Participants) | 13 | 13
units on a scale | -5.3 (4.7) | -5.6 (4.8)

2. Secondary Outcome: Change in Scores in Measurements of Depressive Symptoms (Hamilton Depression Rating Scale, HAM-D), Generalized Anxiety Symptoms (Hamilton Anxiety Rating Scale, HAM-A) and the Sleep Quality Item of the Pittsburgh Sleep Quality Index (PSQI).
Description: Subjects scores on secondary efficacy measures were measured, comparing baseline and the end of 8 weeks of treatment, including the Hamilton Depression Rating Scale, HAM-D, which has 21 items, with scores ranging from 0-66; the Hamilton Anxiety Rating Scale, HAM-A, which has 14 items, with scores ranging from 0-56; and the sleep quality item of the PSQI, a four-point scale rating sleep quality as very good, fairly good, fairly bad or very bad.
Time Frame: Comparing baseline and the end of 8 weeks of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Quetiapine XR | Placebo
Number analyzed (Participants) | 13 | 13
units on a scale
  Decrease in HAM-D scores | 5.0 (5.2) | 3.8 (3.6)
  Decrease in HAM-A scores | 6.8 (8.1) | 5.5 (4.7)
  Increase in PSQI sleep quality scores | 1.3 (0.5) | 1.3 (1.0)

ADVERSE EVENTS:
Groups:
- Quietapine Group: quetiapine SR: Subjects will receive daily dosing at night, with a flexible dosing schedule, 50-400 mg.
- Placebo Group: placebo: Subjects will receive daily dosing at night with caplets matching the appearance of the active drug. However, caplets will not contain any active medication.
Arm/Group | Quietapine Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 10/13 | 5/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quietapine Group (N=13) | Placebo Group (N=13)
Somnolence (Nervous system disorders) | 10 (10) | 5 (5)
Anxiety (Psychiatric disorders) | 4 (4) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1)
Dry Mouth (Nervous system disorders) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 3 (3)
Restlessness (Nervous system disorders) | 2 (2) | 4 (4)
Derealization (Psychiatric disorders) | 2 (2) | 0 (0)
Insomnia (Nervous system disorders) | 1 (1) | 3 (3)
Increased Appetite (Nervous system disorders) | 1 (1) | 2 (2)
Leg Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Weight Loss (Gastrointestinal disorders) | 1 (1) | 0 (0)
Shakiness (Nervous system disorders) | 1 (1) | 0 (0)
Muscle Aches (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Weight Gain (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No